CLINICAL TRIAL: NCT05537259
Title: BUMPP: A Study to Better Understand Mood During the Perinatal Period
Acronym: BUMPP
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: CEHD-2023-31101
Record Dates: First submitted 2022-07-06; First posted 2022-09-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Pregnancy; Postpartum; Mental Health Issue
Keywords: Pregnancy; Postpartum; Mental Health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observation Group: Researchers will collect data on maternal mental health symptoms, as well as health and psychosocial factors, via short interviews (sessions 1 and 4) and via self-report questionnaires completed through REDCap at each session. Participating women will also provide one small hair sample (session 4) for measurement of the stress hormone cortisol and several finger stick blood spot samples (sessions 1,2, and 4) for measurement of immune markers.
  Interventions: Other: Observation Group

INTERVENTIONS:
Other: Observation Group — No intervention; this is an observational study.

SUMMARY:
The overall goal of the BUMPP study is to improve our understanding of a range of moods, feelings, and thoughts that women can experience during pregnancy and soon after they give birth. This study will examine how these moods, feelings, and thoughts are related to changes in hormonal and immune health that women experience during and after pregnancy, and to mother-baby relationships and infant development in the early postpartum months.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* 35 weeks pregnant or less
* carrying only one baby (not twins or triplets)
* first time giving birth
* can speak/read/write in English

Exclusion Criteria:

* major medical health condition like a heart, kidney, or liver disease or HIV
* currently taking corticosteroids, progesterone, or immunosuppressive medications that might impact the samples we are taking in this research study
* have regularly used alcohol, tobacco, or recreational drugs (such as marijuana or prescription drugs for non-medical reasons) during pregnancy (regularly means more than a few times total, such as on a monthly, weekly, or daily basis)

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Pregnant women and their infants
Sampling Method: Non-Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2022-06-27 (Actual); Primary Completion 2023-11-07 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
Self-report questionnaire measure of depressive symptoms (Edinburgh Postnatal Depression Scale) | 35 weeks of pregnancy through 2 months postpartum
  Assessed at each of 4 sessions
Self-report questionnaire measure of anxiety symptoms (Generalized Anxiety Disorder-7) | 35 weeks of pregnancy through 2 months postpartum
  Assessed at each of 4 sessions
Self-report questionnaire measure of manic symptoms (Highs Scale) | 35 weeks of pregnancy through 2 months postpartum
  Assessed at each of 4 sessions
Self-report questionnaire measure of symptoms of psychosis (subscales of Symptom Checklist-90) | 35 weeks of pregnancy through 2 months postpartum
  Assessed at each of 4 sessions
Mother-infant behavior during 5 min play episode coded using Global Rating Scales | 2 months postpartum
  Assessed at in-person laboratory session (session 4)
Bayley Scales of Infant Development, 4th edition, to assess infant cognitive development | 2 months postpartum
  Assessed at in-person laboratory session (session 4)

SECONDARY OUTCOMES:
Monthly cortisol levels determined from hair sample | 35 weeks of pregnancy through 2 months postpartum
  1 sample at session 4
Cytokine levels determined from finger prick blood spot | 35 weeks of pregnancy through 2 months postpartum
  3 samples (sessions 1, 2, and 4)

CONTACTS AND LOCATIONS:
Overall Officials: Megan Gunnar, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States